CLINICAL TRIAL: NCT05589831
Title: Respiratory Support and Brain Health in Preterm Infants: a Prospective Crossover Study
Brief Title: Respiratory Support and Brain Health in Preterm Infants
Status: Recruiting | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 22-0128-A
Record Dates: First submitted 2022-10-05; First posted 2022-10-21 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Sleep; Cerebral Oxygenation
Keywords: Neurally Adjusted Ventilatory Assist; Non-Invasive Positive Pressure Ventilation; Preterm Neonates; Amplitude integrated electroencephalography

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Non-invasive Neurally Adjusted Ventilatory Assist — Neurally Adjusted Ventilatory Assist (NAVA) is a new non-invasive ventilation mode that uses the electrical activity of the diaphragm (EAdi) to offer ventilatory assistance in synchrony with patient effort, thus potentially reducing stress and discomfort. It uses electrodes placed on a modified nasogastric feeding tube to detect the electrical activity of the diaphragm (EAdi), such that both the initiation and termination of a breath during each respiratory cycle is in synchrony with the infant's effort
  Other Names: NIV-NAVA

SUMMARY:
Premature babies often require breathing support during their neonatal intensive care unit stay. This is because their lungs are not fully developed to perform the work of breathing on their own. Although breathing support can be provided via a breathing tube, it is preferable to provide breathing support non-invasively from a breathing machine which is then connected to a mask or prongs placed on the baby's nose. In premature babies born under 32 weeks gestation, a commonly used mode of non-invasive breathing support is called Non-Invasive Positive Pressure Ventilation (NIPPV). In this mode, the breathing machine provides 2 levels of support: one is the constant distending pressure to keep the lungs open and the other provides additional 'breaths' on top of that distending pressure. This is to mimic regular breathing. These breaths are set at a fixed rate and pressure. Although NIPPV protects the lungs from injury caused by a breathing tube, the breaths are not in sync with the baby's own breathing effort. Another mode of non-invasive breathing support recently being used in premature infants called Neurally Adjusted Ventilatory Assist (NAVA). When NAVA is provided non-invasively using a mask or prongs similar to NIPPV, it is called Non-invasive NAVA (NIV-NAVA). During NIV-NAVA a special feeding tube is used that detects the baby's own breathing movement from the electrical signal of the baby's diaphragm and feeds back to the machine which then provides a 'top-up' to the baby's own breath. This top-up breath also provides only as much pressure as the baby needs on top on their own breathing effort. Therefore, this is thought to be in sync with the baby's own breathing effort. However, it is not known if this mode of ventilation leads to improved sleep, improved brain oxygen levels, reduced discomfort and improved functioning of the diaphragm. The investigators aim to examine these indices in this research project.

DETAILED DESCRIPTION:
Rationale: It is imperative to find the optimal method of supporting not only lung development, but also brain development during this critical period of brain growth and development. NIV-NAVA is a more physiologically compatible method of supporting respiration. The investigators hypothesize that this compatibility may increase comfort and restful periods compared to standard NIPPV, and thus, may be more neuroprotective.

Objective and outcomes assessed: The objective is to compare sleep-wake cycling, cerebral oxygenation, heart rate variability and diaphragm function during standard NIPPV and NIV-NAVA modes in preterm neonates born at <32 weeks' gestation who are stable on NIPPV or NIV-NAVA for at least 24 hours and are a minimum of 3 days old.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born between 22+0 and 31+6 weeks' GA
* Weight > 500 g at the time of approach for consent
* A minimum of 3 days of age
* Clinically stable for > 24 hours while receiving NIPPV or NIV-NAVA

Clinical stability will be defined as meeting all the following criteria for a 24 hour period prior to recruitment:

1. differences in maximum and minimum fractions of inspired oxygen (FiO2) of <20%
2. differences in maximum and minimum MAP <4 cm H2O
3. no active infection
4. no hypotension
5. no use of cardioactive medications or medical therapy for patent ductus arteriosus.

Exclusion Criteria:

* Infants with IVH of grade 3 or 4
* Birth weight < 3rd percentile
* Genetic or congenital abnormalities

Min Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Preterm infants at tertiary NICU at Mount Sinai Hospital (Toronto, Ontario).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of uninterrupted sleep-wake cycling (SWC) | For 24 hours after intervention initiation
  An uninterrupted SWC will be defined as a smooth and gradual decrease in the minimum amplitude on aEEG to quiet sleep (QS), followed by a gradual increase to active sleep or awake state (AS). An interrupted SWC will be defined as a sudden or sharp increase in the minimum amplitude during QS with change to AS state that may or may not be followed by a further drop in QS.

SECONDARY OUTCOMES:
Total duration of quiet sleep (QS) | For 24 hours after intervention initiation
  First, high base voltage (HBV) will be defined as the voltage of the lower margin of aEEG during AS. Total QS duration will be calculated as the combined duration of time spent below the HBV in uninterrupted SWC during 24 h.
Cerebral oxygen saturation (CrSO2) | For 24 hours after intervention initiation
  Cerebral fractional tissue oxygen extraction (CFTOE), calculated as (oxygen saturation [SpO2] - CrSO2) / SpO2, will be calculated offline
Newborn Infant Parasympathetic Evaluation (NIPE) index | For 24 hours after intervention initiation
  Measurement of heart rate variability
Diaphragmatic thickness | 1 day during Nasal Intermittent Positive-Pressure Ventilation (NIPPV) period and 1 day during the Non-Invasive Neurally Adjusted Ventilatory Assist (NIV-NAVA) period
  Measurement of Diaphragmatic thickness (DT) using lung ultrasound
Diaphragm thickness fraction | 1 day during Nasal Intermittent Positive-Pressure Ventilation (NIPPV) period and 1 day during the Non-Invasive Neurally Adjusted Ventilatory Assist (NIV-NAVA) period
  Diaphragmatic thickness fraction (DTF), calculated as ([(inspiratory thickness-expiratory thickness)]) / (expiratory thickness) x 100, will be calculated using diaphragmatic thicknesses obtained from lung ultrasound
Diaphragmatic excursion (DE) | 1 day during Nasal Intermittent Positive-Pressure Ventilation (NIPPV) period and 1 day during the Non-Invasive Neurally Adjusted Ventilatory Assist (NIV-NAVA) period
  Measurement of Diaphragmatic excursion (DE) using lung ultrasound
Lung Ultrasound Severity Score (LUSS) | 1 day during Nasal Intermittent Positive-Pressure Ventilation (NIPPV) period and 1 day during the Non-Invasive Neurally Adjusted Ventilatory Assist (NIV-NAVA) period
  Point score based on qualitative analysis using lung ultrasound. For each lung area, a 0- to 3-point score is given. Where 0 score refer to normal aeration and 3 score refer to severe loss of lung aeration. Total score ranging from 0-18 based on 3 areas on each lung, with low score means good lung aeration and higher means poor lung aeration.

CONTACTS AND LOCATIONS:
Overall Officials: Poorva Deshpande, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No